CLINICAL TRIAL: NCT04796610
Title: Mopati: A Pilot Hiv Treatment Partner Intervention In Botswana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other); Children's Mercy Hospital Kansas City (Other); University of Botswana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH121229 (NIH)
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: HIV
Keywords: HIV; Treatment partner

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention patients (Experimental): Unsuppressed HIV patients at the intervention clinic will receive guidance from their health care provider on the selection of a treatment partner. The patient will receive education on HIV treatment and how treatment partners can support patients in treatment adherence.
  Interventions: Behavioral: Mopati
- Control patients (No Intervention): Patients at the control clinic will receive standard of care at the clinic during the intervention assessment period.
- Intervention treatment partners (Experimental): Unsuppressed HIV patients at the intervention clinic will receive guidance from their health care provider on the selection of a treatment partner. The treatment partner will receive education on HIV treatment and how treatment partners can support patients in treatment adherence.
  Interventions: Behavioral: Mopati
- Control treatment partners (No Intervention): Treatment partners will not receive any intervention; treatment partners' patients at the control clinic will receive standard of care at the clinic during the intervention assessment period.

INTERVENTIONS:
Behavioral: Mopati — The intervention will provide training to health care providers on how to guide unsuppressed HIV patients in the selection of treatment partners. The Mopati program will provide education to patients and their treatment partners about HIV treatment and how treatment partners can support patients in treatment adherence.
  Arms: Intervention patients; Intervention treatment partners

SUMMARY:
This study is a pilot test of the Mopati program ("partner" in Setswana), which is a multi-level intervention that guides healthcare providers and patients about treatment partner selection, and trains treatment partners on provision of effective support. The Specific Aims are: (1) To develop a multi-level treatment partner intervention with input from community and healthcare provider stakeholders in Botswana; and (2) To conduct a pilot test of the feasibility, acceptability, and preliminary effects on viral suppression.

DETAILED DESCRIPTION:
This study will train health care providers to guide unsuppressed HIV positive patients in the selection of a treatment partner. All health care providers at the intervention clinic (e.g., physicians, nurses, peer counselors) will be educated about effective characteristics of treatment partners, and provided with standard guidance about treatment partner selection to deliver to all patients initiating ART or who are not suppressed (however, for increased impact, the investigators will test the intervention only among those not suppressed). The standard guidance will incorporate Motivational Interviewing (MI) strategies, to acknowledge patients' difficulties and offer advice without trying to force the patient to select a treatment partner of a particular type.

The intervention clinic will sponsor group sessions for treatment partners of unsuppressed patients, to educate treatment partners about HIV treatment, and train treatment partners on counseling skills to convey acceptance of and compassion, and to be non-judgmental and non-confrontational. The investigators will train treatment partners in core MI skills of open questions and reflective listening, to avoid confrontations and support patients in developing motivation for adherence. In the training, the investigators will use experiential learning methods to help partners to understand that confronting their partners about poor adherence, while born out of love and concern for patients' health, is ineffective. The investigators do not intend for treatment partners to be proficient in all MI counseling strategies, but the investigators will train treatment partners to use the two core MI skills. Patients and their treatment partners will be asked to attend at least 3 sessions over the 3-month intervention period. The investigators will survey patients and treatment partners at baseline and 3-months post-baseline and collect viral load from clinic records. Intervention feasibility and acceptability will be assessed via mixed methods (e.g., semi- structured interviews with patients, treatment partners, and clinic staff; refusal rates).

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they are: 1) 18 years of age or older, 2) On antiretroviral treatment for HIV (ART) and initiated ART at least 6 months prior, and 3 ) Not virally suppressed (one viral load ≥ 400 cp/ml within prior 12 months at time of enrollment).
* Treatment partners will be eligible if they are 18 years of age or older and selected to be a patient's treatment partner.

Exclusion Criteria:

* Patients will not be eligible if they screen positive for HIV-related dementia or if they show ART resistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bogart, PhD, Principal Investigator — RAND; Mosepele Mosepele, MD, MPH, Principal Investigator — University of Botswana & Botswana Harvard AIDS Institute Partnership
Locations (1):
- Botswana Harvard AIDS Institute Partnership (BHP), Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bogart LM, Phaladze N, Kgotlaetsile K, Klein DJ, Goggin K, Mosepele M. Pilot Test of Mopati, a Multi-Level Adherence Intervention for People Living with HIV and Their Treatment Partners in Botswana. Int J Behav Med. 2024 Oct;31(5):787-798. doi: 10.1007/s12529-023-10233-7. Epub 2023 Nov 13. PMID 37957535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note that both patients and treatment partners were recruited and participated in the intervention. However, results are only reported for patients (and not treatment partners) as the primary and secondary trial outcomes apply to patients only.
Pre-assignment Details: COVID-19 was a large challenge to recruitment and study implementation as a whole
Groups:
- Intervention Patients; Intervention Treatment Partners: Unsuppressed patients with HIV at the intervention clinic will receive guidance from their health care provider on the selection of a treatment partner. The patient and treatment partner will receive education on HIV treatment and how treatment partners can support patients in treatment adherence.
- Control Treatment Partners: Treatment partners of patients at the control clinic who will receive standard of care at the clinic during the intervention assessment period.
Period: Overall Study
Arm/Group | Intervention Patients | Control Patients | Intervention Treatment Partners | Control Treatment Partners
Started | 30 | 30 | 17 | 28
Completed | 27 | 30 | 16 | 27
Not Completed | 3 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 30 patients in the intervention clinic and 30 patients in the control clinic
Groups:
- Intervention Patients: Unsuppressed HIV patients at the intervention clinic will receive guidance from their health care provider on the selection of a treatment partner. The patient and treatment partner will receive education on HIV treatment and how treatment partners can support patients in treatment adherence.
  The Mopati intervention provides (1) training to health care providers on how to guide unsuppressed HIV patients in the selection of treatment partners and (2) education to patients and their treatment partners about HIV treatment and how treatment partners can support patients in treatment adherence.
  Note that both patients and treatment partners were recruited and participated in the intervention. However, counts, baseline characteristics, and results are only reported for patients (and not treatment partners) as the primary and secondary trial outcomes apply to patients only.
- Intervention Treatment Partners: Unsuppressed HIV patients at the intervention clinic will receive guidance from their health care provider on the selection of a treatment partner. The patient and treatment partner will receive education on HIV treatment and how treatment partners can support patients in treatment adherence.
- Total: Total of all reporting groups
Arm/Group | Intervention Patients | Control Patients | Intervention Treatment Partners | Control Treatment Partners | Total
Number analyzed (Participants) | 30 | 30 | 17 | 28 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (10.4) | 43.8 (11.6) | 40.8 (11.2) | 40.1 (9.5) | 40.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 12 | 22 | 71
  Male | 12 | 11 | 5 | 6 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 30 | 30 | 17 | 28 | 105
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Botswana | 30 | 30 | 17 | 28 | 105
Viral Suppression [Count of Participants; unit: Participants] — Population: Patients were not virally suppressed at baseline per eligibility criteria. Treatment partner viral suppression data was not collected from medical records as was done for patients. Note that treatment partners did not have to be HIV-positive to be eligible.
  Participants
    number analyzed (Participants) | 30 | 30 | 0 | 0 | 60
    (all) | 0 | 0 | 0 | 0 | 0
Self-reported Adherence [Count of Participants; unit: Participants] — Adherence measured as self-reported percentage of doses taken in last month, dichotomized as at least 95% of doses taken in last month Population: 2 intervention patients did not complete the baseline survey and could not be reached after multiple attempts. One control patient declined to respond to this item.
  Treatment partner adherence was asked only of treatment partners who were HIV-positive (treatment partners did not have to be HIV-positive to be eligible.) One HIV-positive control treatment partner and one HIV-positive intervention treatment partner declined to respond to this item.
  Participants
    number analyzed (Participants) | 28 | 29 | 7 | 11 | 75
    (all) | 18 | 23 | 6 | 10 | 57
Non-Directive Support [Mean (Standard Deviation); unit: units on a scale] — Patient perceptions of non-directive support (α = .92) from their treatment partner were assessed with a subscale adapted from the Social Support Inventory. Response options were 1, "not at all typical" to 5, "very typical." Higher values were indicative of greater non-directive support. Population: 2 intervention patients did not complete baseline survey and could not be reached after multiple attempts. An additional 3 intervention patients declined to respond to this item.
  Treatment partner non-directive support was only asked of the N=15 treatment partners who were (a) HIV-positive and (b) reported that the patient is also their treatment partner.
  units on a scale
    number analyzed (Participants) | 25 | 30 | 3 | 12 | 70
    (all) | 4.4 (1.0) | 4.6 (0.7) | 4.8 (0.3) | 4.8 (0.7) | 4.6 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Viral Suppression of Patient Participants
Description: Viral suppression will be defined as viral load < 400 cp/ml
Time Frame: 6 months
Population: Viral load was collected from medical records of previous clinic visits. Viral load was only used in analysis if the participant had a viral load measurement between 90 and 180 days after the baseline survey and, if an intervention participant, after the last intervention session. Because medical records often did not include a viral load measurement in the required date range, viral suppression was not available for all participants.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Patients: Unsuppressed HIV patients at the intervention clinic will receive guidance from their health care provider on the selection of a treatment partner. The patient and treatment partner will receive education on HIV treatment and how treatment partners can support patients in treatment adherence.
  Mopati: The intervention will provide training to health care providers on how to guide unsuppressed HIV patients in the selection of treatment partners. The Mopati program will provide education to patients and their treatment partners about HIV treatment and how treatment partners can support patients in treatment adherence.
Arm/Group | Intervention Patients | Control Patients
Number analyzed (Participants) | 18 | 16
Participants | 12 | 13
Statistical Analysis 1: Comparison: Intervention Patients vs Control Patients; Test type: Superiority; p = 0.49, Regression, Logistic; Model is adjusted for participant age; Odds Ratio (OR) = .55, 95% CI 2-sided [.1 to 2.98] — Results are presented for an indicator where 0=control and 1=intervention

2. Secondary Outcome: Number of Patient Participants Self-Reported as Treatment Adherent
Description: Participants self-reported the percentage of doses taken in the past month; we defined treatment adherence as having taken at least 95% of prescribed doses
Time Frame: 3-months post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Patients | Control Patients
Number analyzed (Participants) | 27 | 30
Participants | 24 | 22
Statistical Analysis 1: Comparison: Intervention Patients vs Control Patients; Test type: Superiority; p = .011, Regression, Logistic — Model is adjusted for participant age; Odds Ratio (OR) = 16.82, 95% CI 2-sided [1.93 to 146.91] — Results are presented for an indicator where 0=control and 1=intervention

3. Secondary Outcome: Perceived Treatment Partner Support
Description: Continuous scores on Nondirective Support scale (0-5); higher = more nondirective support, rated by patient participants
Time Frame: 3-months post-baseline
Population: Some participants skipped the scale on the survey assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Patients | Control Patients
Number analyzed (Participants) | 21 | 30
units on a scale | 4.9 (0.2) | 4.5 (1.0)
Statistical Analysis 1: Comparison: Intervention Patients vs Control Patients; Test type: Superiority; p = .03, Regression, Linear; Model is adjusted for participant age; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.07 to 0.97] — Results are presented for an indicator where 0=control and 1=intervention

ADVERSE EVENTS:
Time Frame: 3 months
Description: The definition was similar as the clinicaltrials.gov definition, and additionally included systematic assessment of current intimate partner violence
Groups:
- Intervention: Unsuppressed patients with HIV at the intervention clinic will receive guidance from their health care provider on the selection of a treatment partner. The patient and treatment partner will receive education on HIV treatment and how treatment partners can support patients in treatment adherence.
- Control: Patients at the control clinic will receive standard of care at the clinic during the intervention assessment period.
- Intervention - Treatment Partners: Treatment partners of unsuppressed patients with HIV at the intervention clinic received education on HIV treatment and how treatment partners can support patients in treatment adherence.
- Control - Treatment Partners: Treatment partners of unsuppressed patients with HIV at the control clinic did not receive any intervention.
Arm/Group | Intervention | Control | Intervention - Treatment Partners | Control - Treatment Partners
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/17 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/17 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/17 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04796610/Prot_SAP_000.pdf